CLINICAL TRIAL: NCT01309243
Title: A Phase 3B, Randomized, Open-label Study to Evaluate the Safety and Efficacy of a Single Tablet Regimen of Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate Compared With a Single Tablet Regimen of Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Brief Title: Study to Evaluate the Safety and Efficacy of a Single Tablet Regimen of Emtricitabine/Rilpivirine/Tenofovir Disoproxil Fumarate Compared With a Single Tablet Regimen of Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in HIV-1 Infected, Antiretroviral Treatment-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-264-0110
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: HIV-1 Infection
Keywords: HIV; HIV-1; Antiretroviral Treatment-Naïve
MeSH Terms: interventions — Emtricitabine, Rilpivirine, Tenofovir Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTC/RPV/TDF (Experimental)
  Interventions: Drug: FTC/RPV/TDF
- EFV/FTC/TDF (Experimental)
  Interventions: Drug: EFV/FTC/TDF

INTERVENTIONS:
Drug: FTC/RPV/TDF — Emtricitabine (FTC) 200 mg/rilpivirine (RPV) 25 mg/tenofovir disoproxil fumarate (TDF) 300 mg single-tablet regimen administered orally once daily with a meal
  Other Names: Complera®; Eviplera®
  Arms: FTC/RPV/TDF
Drug: EFV/FTC/TDF — Efavirenz (EFV) 600 mg/FTC 200 mg/TDF 300 mg single-tablet regimen administered orally once daily on an empty stomach, preferably at bedtime
  Other Names: Atripla®
  Arms: EFV/FTC/TDF

SUMMARY:
The purpose of the study was to evaluate the safety and efficacy of the emtricitabine (FTC)/rilpivirine (RPV)/tenofovir disoproxil fumarate (TDF) single-tablet regimen (STR) compared with the efavirenz (EFV)/FTC/TDF STR in HIV-1 infected adults who had not previously received treatment with antiretroviral medications.

Participants were randomized in a 1:1 ratio to receive one of the study treatments. Randomization was stratified by HIV-1 RNA level (≤ 100,000 copies/mL or > 100,000 copies/mL) at screening. A treatment duration of 96 weeks was planned, with the option for subjects in FTC/RPV/TDF STR arm to receive treatment following the Week 96 visit until FTC/RPV/TDF STR is commercially available or until Gilead Sciences elects to terminate development in that country.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign a written informed consent form
* Plasma HIV-1 RNA levels ≥ 2,500 copies/mL at screening
* No prior use of any approved or experimental anti-HIV drug for any length of time
* Screening genotype report showing sensitivity to EFV, FTC, TDF, and lack of the RPV mutations K101E/P, E138A/G/K/Q/R, Y181C/I/V, and H221Y
* Normal ECG
* Hepatic transaminases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) ≤ 5 x the upper limit of the normal range (ULN)
* Total bilirubin ≤ 1.5 mg/dL, or normal direct bilirubin
* Adequate hematologic function
* Serum amylase ≤ 5 x ULN (participants with serum amylase > 5 x ULN remained eligible if serum lipase was ≤ 5 x ULN)
* Adequate renal function
* Males and Females of childbearing potential must have agreed to utilize highly effective contraception methods (two separate forms of contraception, one of which must be an effective barrier method, or be non-heterosexually active, practice sexual abstinence or have a vasectomized partner) from screening throughout the duration of study period and for 12 weeks following the last dose of study drug.
* Adult (≥ 18 years) males or non-pregnant females

Exclusion Criteria:

* A new AIDS-defining condition diagnosed within the 30 days prior to screening
* Females who were breastfeeding
* Positive serum pregnancy test (female of childbearing potential)
* Proven or suspected acute hepatitis in the 30 days prior to study entry
* Subjects receiving drug treatment for hepatitis C, or subjects who were anticipated to receive treatment for hepatitis C during the course of the study
* Subjects experiencing decompensated cirrhosis
* Had an implanted defibrillator or pacemaker
* Current alcohol or substance abuse
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous carcinoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to baseline
* Receiving ongoing therapy or anticipated to need to initiate drugs or herbal/natural supplements during the study that are contraindicated or not recommended for use, including drugs not to be used with FTC, EFV, RPV, or TDF; or subjects with known allergies to the excipients of the FTC/RPV/TDF or EFV/FTC/TDF single-tablet regimens
* Participation in any other clinical trial without prior approval from the sponsor was prohibited while participating in this trial.
* Had been treated with immunosuppressant therapies or chemotherapeutic agents within 3 months of study screening, or expected to receive these agents or systemic steroids for immunosuppression during the study (eg, corticosteroids, immunoglobulins, and other immune-based or cytokine-based therapies)
* Had any other clinical condition or prior therapy that, in the opinion of the Investigator, would have made the participant unsuitable for the study or unable to comply with the dosing requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Fralich, M.D., Study Chair — Gilead Sciences
Locations (151):
- United States (83):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Spectrum Medical Group, Phoenix, Arizona
  - AHF Research Center, Beverly Hills, California
  - Kaiser Permanente Medical Center, Hayward, California
  - Living Hope Education and Research Consultants, Long Beach, California
  - Kaiser Permanente Medical Center, Los Angeles, California
  - Jeffrey Goodman Special Care Clinic/Los Angeles Gay and Lesbian Center, Los Angeles, California
  - Lightsource Medical, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Oasis Clinic, Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Orange Coast Medical Group, Newport Beach, California
  - East Bay AIDS Center, Oakland, California
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical/Dr.Fritz, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, San Francisco, California
  - Apex Research LLC, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Clinic, Washington D.C., District of Columbia
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - Medical Faculty Associates, Washington D.C., District of Columbia
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Gary J. Richmond, M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - The Kinder Medical Group, Miami, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Valuhealthmd,Llc / Idocf, Orlando, Florida
  - Infectious Disease Associates of NW FL, Pensacola, Florida
  - AHF Health Positive - Tampa Bay, Safety Harbor, Florida
  - St. Joseph's Hospital d/b/a Comprehensive Research Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Atlanta ID Group, Atlanta, Georgia
  - Infectious Disease Specialists of America, Decatur, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - Clint Spencer Clinic, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - Johns Hopkins Rockland Physicians Practice and Research Group at Greenspring Station, Lutherville, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Claudia T Martorell, MD., LLC dba The Research Institute, Springfield, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Central West Clinical Research, Inc., St Louis, Missouri
  - Southampton Healthcare, St Louis, Missouri
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Southwest Care Center, Sante Fe, New Mexico
  - Upstate Infectious Disease Associates, Albany, New York
  - New York Hospital Queens, Flushing, New York
  - North Shore University Hospital--Division of Infectious Diseases, Manhasset, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - Ricky K. Hsu, Md, Pc, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Clinical and Translational Research Center - UNC Hospitals, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - Rosedale Infectious Diseases, Huntersville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System Care Center, Akron, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - University of South Carolina, Columbia, South Carolina
  - Central Texas Clinical Research, Austin, Texas
  - Trinity Health and Wellness Center, Dallas, Texas
  - Southwest Infectious Disease Associates, Inc., Dallas, Texas
  - Tarrant County Infectious Disease Associates, Fort Worth, Texas
  - Garcia Family Health Group, Harlingen, Texas
  - Therapeutic Concepts, P.A., Houston, Texas
  - Gordon E. Crofoot MD PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - CARE-ID, Annandale, Virginia
  - Peter Shalit, M.D., Seattle, Washington
  - Rockwood Pulmonary and Critical Care, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (8):
  - Holdsworth House Medical Practice, Darlinghurst, New South Wales
  - St Vincent's Hospital, Sydney, Darlinghurst
  - Taylor Square Private Clinic, Darlinghurst
  - Northside Clinic, Fitzroy North
  - Clinical Research - Infectious Diseases Unit Alfred Hospital, Melbourne
  - Prahran Market Clinic, Prahran
  - Albion Street Centre, Surry Hills
  - East Sydney Doctors, Sydney
- Austria (3):
  - LKH Medical University Graz West, Department of Internal Medicine, Graz
  - Universitätsklinikum Innsbruck Universitätsklinik für Dermatologie und Venerologie, Innsbruck
  - Department of Dermatology, Allergy, and Infectious Disease University Vienna Medical School, Vienna
- Belgium (3):
  - Institute of Tropical Medicine, Antwerp
  - Cliniques Universitaires Saint-Luc - UCL, Brussels
  - University Hospitals Leuven, Leuven
- Canada (8):
  - Division of HIV/AIDS, St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Maple Leaf Research Maple Leaf Medical Clinic, Toronto, Ontario
  - University Health Network/Toronto General Hospital, Toronto, Ontario
  - Clinique médicale L' Actuel, Montreal, Quebec
  - McGill University Health Center, Montreal Chest Institute, Montreal, Quebec
- France (10):
  - Hopital Raymond Poincare, Garches
  - Hôpital de la Croix-Rousse, Lyon
  - Chu Hotel Dieu, Nantes
  - CHU Nice - Archet 1, Nice
  - Hopital Bichat Claude Bernard, Paris
  - HOSPITAL SAINT LOUIS - Services des Maladies Infectieuses, Paris
  - Hopital Saint Antoine- Service Maladies infectieuses, Paris
  - Hôpital Pitié Salpêtrière - Service des Maladies Infectieuses, Paris
  - Hopital Tenon Service des Maladies infectieuses et tropicales, Paris
  - Centre Hospitalier de Tourcoing, Tourcoing
- Germany (8):
  - EPIMED GmbH, Berlin
  - Medizinische Universitätsklinik I der Friedrich-Wilhelms Universität Bonn, Bonn
  - Department of Dermatology University Hospital Essen, Essen
  - Private Practice Gute & Locher & Lutz, Infektiologikum, Frankfurt am Main
  - Division of Infectious Disease, Department of Medicine, University Hospital Freiburg, Freiburg im Breisgau
  - ICH Study Center, Hamburg
  - Universitätsklinikum Eppendorf Ambulanzzentrum des UKE GmbH, Infekiologie, Hamburg
  - MUC Research GmbH, München
- Italy (6):
  - Ospedali Riuniti, Bergamo
  - IRCCS Ospedale San Raffaele Centro San Luigi, Unità Operativa di Malattie Infettive, Milan
  - I Div Infectious Diseases, Luigi Sacco Hospital, Milan
  - San Gerardo Hospital - Uo Malattie Infettive, Monza
  - Foundation "IRCCS Policlinico San Matteo Hospital", Pavia
  - National Institute for Infectious Diseases "L. Spallanzani" IRCCS, Rome
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Erasmus MC, Rotterdam
- Portugal (3):
  - Hospital de Santa Maria - CHLN, EPE, Lisbon
  - Serviço de Doenças Infecciosas, Hospital S. Joao, Porto
  - Hospital de Joaquim urbano, Porto
- Clinical Research Puerto Rico, San Juan, Puerto Rico
- Spain (6):
  - Hospital General Universitario Alicante, Alicante
  - Hospital Universitari de Bellvitge, Cataluña
  - Hospital Universitario de Elche, Unidad de Enfermedades Infecciosas, Elche
  - Hospital Universitario 12 Octubre, Madrid
  - Unidad HIV. Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
- Switzerland (3):
  - Universitätsklinik für Infektiologie, Bern
  - CHUV, Lausanne
  - University Hospital Zurich, Zurich
- United Kingdom (7):
  - Royal Sussex County Hospital, Brighton
  - Ridu, Wgh, Edinburgh
  - Clinical Research, Grahame Hayton Unit Ambrose King Centre, The Royal London Hospital, London
  - Royal Free NHS Trust,, London
  - Guys and St Thomas' NHS trust, London
  - Chelsea and Westminster Hospital, London
  - North Manchester General Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in a total of 121 study sites in North America, Europe, and Australia. The first participant was screened on 23 February 2011. The last participant observation was on 03 February 2014.
Pre-assignment Details: 991 participants were screened.
Groups:
- FTC/RPV/TDF: Emtricitabine (FTC) 200 mg/rilpivirine (RPV) 25 mg/tenofovir disoproxil fumarate (TDF) 300 mg single-tablet regimen (STR) administered orally once daily
- EFV/FTC/TDF: Efavirenz (EFV) 600 mg/FTC 200 mg/TDF 300 mg STR administered orally once daily
Period: Randomized Phase Through Week 96
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Started | 400 | 399
Randomized and Treated | 394 | 392
Completed | 316 | 290
Not Completed | 84 | 109
Not completed — Randomized but not treated | 6 | 7
Not completed — Adverse Event | 12 | 43
Not completed — Death | 0 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Lack of Efficacy | 16 | 4
Not completed — Investigators Discretion | 3 | 6
Not completed — Withdrew Consent | 12 | 18
Not completed — Lost to Follow-up | 23 | 22
Not completed — Subject Non-Compliance | 9 | 7
Not completed — Protocol Violation | 1 | 1
Period: Extension Phase
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Started | 40 (40 participants from the Randomized Phase continued the study in the Extension Phase.) | 117 (117 participants from the Randomized Phase continued the study in the Extension Phase.)
Completed | 34 | 117
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the Safety Analysis Set (randomized and received at least 1 dose of study drug) were analyzed for baseline characteristics.
Groups:
- FTC/RPV/TDF: FTC 200 mg/RPV 25 mg/TDF 300 mg STR administered orally once daily
- EFV/FTC/TDF: EFV 600 mg/FTC 200 mg/TDF 300 mg STR administered orally once daily
- Total: Total of all reporting groups
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF | Total
Number analyzed (Participants) | 394 | 392 | 786
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (10.4) | 37 (11.0) | 37 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 366 | 364 | 730
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 8 | 13 | 21
  Black or African Heritage | 98 | 94 | 192
  Native Hawaiian or Pacific Islander | 4 | 3 | 7
  White | 266 | 262 | 528
  Other | 13 | 19 | 32
  Not Permitted | 1 | 0 | 1
  Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 59 | 75 | 134
  Non-Hispanic/Latino | 331 | 315 | 646
  Not Permitted | 3 | 2 | 5
  Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for Region of Enrollment
  participants
    United States | 262 | 279 | 541
    Australia | 15 | 25 | 40
    Canada | 28 | 20 | 48
    Germany | 25 | 22 | 47
    France | 16 | 7 | 23
    United Kingdom | 12 | 8 | 20
    Puerto Rico | 8 | 10 | 18
    Spain | 9 | 6 | 15
    Italy | 10 | 3 | 13
    Belgium | 4 | 5 | 9
    Portugal | 2 | 5 | 7
    Switzerland | 2 | 3 | 5
    Austria | 7 | 6 | 13
HIV-1 RNA [Mean (Standard Deviation); unit: log10 copies/mL] | 4.8 (0.65) | 4.8 (0.61) | 4.8 (0.63)
HIV-1 RNA Category [Number; unit: participants]
  ≤ 100,000 copies/mL | 260 | 250 | 510
  > 100,000 copies/mL | 134 | 142 | 276
Cluster of differentiation 4 (CD4) Cell Count [Mean (Standard Deviation); unit: cells/μL] | 395.7 (179.64) | 385.2 (186.82) | 390.5 (183.21)
Use of lipid-lowering agent [Number; unit: participants]
  Yes | 4 | 1 | 5
  No | 390 | 391 | 781

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the US FDA snapshot algorithm.
  The snapshot algorithm defines a patient's virologic response status using only the viral load at the predefined time point within an allowed window of time.
Time Frame: Week 48
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 394 | 392
percentage of participants | 85.8 | 81.6
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; The analysis was to assess the noninferiority of FTC/RPV/TDF versus EFV/FTC/TDF using a 95% confidence interval (CI) approach, with a noninferiority margin of 12% (lower bound of CI > -12%). 700 subjects allocated 1:1 to either treatment arm was predicted to give > 95% power when the proportion of responders in both treatment groups for the primary endpoint is 80% at Week 48; Test type: Non-Inferiority or Equivalence — Null hypothesis: The FTC/RPV/TDF group was at least 12% worse than the EFV/FTC/TDF group with respect to the percentage of subjects achieving HIV-1 RNA < 50 copies/mL ("response rate," as defined by the snapshot analysis algorithm) at Week 48. Alternative hypothesis: The FTC/RPV/TDF group was less than 12% worse than the EFV/FTC/TDF group with respect to the percentage of subjects achieving HIV-1 RNA < 50 copies/mL at Week 48; Difference in the response rates = 4.1, 95% CI 2-sided [-1.1 to 9.2] — The baseline stratum-weighted (HIV-1 RNA ≤ 100,000 and > 100,000 copies/mL) difference in virologic success rates and its 95% CI were from baseline HIV-1 RNA adjusted Mantel-Haenszel proportions

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the US FDA snapshot algorithm.
Time Frame: Baseline to Week 96
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 394 | 392
percentage of participants | 77.9 | 72.4
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; Difference in the response rates = 5.5, 95% CI 2-sided [-0.6 to 11.5] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Full Analysis Set with available data were analyzed; the missing = excluded method was used in which all participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 357 | 346
cells/μL | 200 (158.6) | 191 (144.3)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p = 0.34, ANOVA — The p-value, and difference in least square means (LSM) and its 95% CI are from analysis of variance (ANOVA) with treatment and baseline HIV-1 RNA levels (≤ 100,000, > 100,000 copies/mL) as fixed effect; Difference in LSM = 11, 95% CI 2-sided [-11 to 32]

4. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline to Week 96
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 327 | 319
cells/μL | 278 (186.6) | 259 (191.4)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p = 0.17, ANOVA — The p-value, and difference in LSM and its 95% CI are from ANOVA with treatment and baseline HIV-1 RNA levels (≤ 100,000, > 100,000 copies/mL) as fixed effect; Difference in LSM = 20, 95% CI 2-sided [-9 to 49]

5. Secondary Outcome: Change From Baseline in Fasting Total Cholesterol at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed using the missing = excluded method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 322 | 305
mg/dL | 1 (28.1) | 22 (31.3)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for the difference in change from baseline at Week 48 is from ANOVA with treatment as fixed effect

6. Secondary Outcome: Change From Baseline in Fasting High-density Lipoprotein (HDL) Cholesterol at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed using the missing = excluded method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 322 | 305
mg/dL | 2 (8.7) | 8 (10.3)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for the difference in change from baseline at Week 48 is from ANOVA with treatment as fixed effect

7. Secondary Outcome: Change From Baseline in Fasting Low-density Lipoprotein (LDL) Cholesterol at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed using the missing = excluded method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 322 | 303
mg/dL | 1 (24.4) | 14 (28.2)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for the difference in change from baseline at Week 48 is from ANOVA with treatment as fixed effect

8. Secondary Outcome: Change From Baseline in Fasting Triglycerides at Week 48
Time Frame: Baseline to Week 48
Population: Participants in the Safety Analysis Set with available data were analyzed using the missing = excluded method.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 322 | 305
mg/dL | -8 (68.9) | 8 (103.0)
Statistical Analysis 1: Comparison: FTC/RPV/TDF vs EFV/FTC/TDF; Test type: Superiority or Other; p < 0.001, ANOVA — P-value for the difference in change from baseline at Week 48 is from ANOVA with treatment as fixed effect

9. Secondary Outcome: Development of HIV-1 Drug Resistance Through Week 96, All Participants
Description: Participants who experienced either suboptimal virologic response or virologic rebound were considered to have virologic failure and were analyzed for resistance. Suboptimal virologic response was assessed at Week 8 and was defined as having HIV-1 RNA ≥ 50 copies/mL and < 1-log10 reduction from baseline at the Week 8 visit, which was confirmed at the subsequent visit. Virologic rebound was defined as having 2 consecutive visits with HIV-1 RNA ≥ 400 copies/mL after achieving HIV-1 RNA < 50 copies/mL, or as having 2 consecutive visits with > 1 log10 increase in HIV-1 RNA from their nadir. In addition, subjects who were on study drugs, had not been analyzed previously, and who had HIV-1 RNA ≥ 400 copies/mL at Week 48, Week 96, or their last visit (at or after Week 8) were also analyzed for resistance at their last visit. Subsequent to the first resistance testing, subjects experiencing repeated confirmed virologic failure were assessed for resistance retesting on a case-by-case basis.
Time Frame: Baseline to Week 96
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 394 | 392
percentage of participants
  Baseline through Week 48 | 4.3 | 0.8
  Week 48 through Week 96 | 1.0 | 0.3
  Baseline through Week 96 | 5.3 | 1.0

10. Secondary Outcome: Development of HIV-1 Drug Resistance Through Week 96, Participants With Viral Resistance
Description: Resistance Analysis Set: participants with either suboptimal virologic response or virologic rebound were considered to have virologic failure and were analyzed. Suboptimal virologic response was assessed at Week 8 and was defined as having HIV-1 RNA ≥ 50 copies/mL and < 1-log10 reduction from baseline at the Week 8 visit, which was confirmed at the subsequent visit. Virologic rebound was defined as having 2 consecutive visits with HIV-1 RNA ≥ 400 copies/mL after achieving HIV-1 RNA < 50 copies/mL, or as having 2 consecutive visits with > 1 log10 increase in HIV-1 RNA from their nadir. In addition, subjects who were on study drugs, had not been analyzed previously, and who had HIV-1 RNA ≥ 400 copies/mL at Week 48, Week 96, or their last visit (at or after Week 8) were also analyzed for resistance at their last visit. Subsequent to the first resistance testing, subjects experiencing repeated confirmed virologic failure were assessed for resistance retesting on a case-by-case basis.
Time Frame: Baseline to Week 96
Population: Resistance Analysis Set
Measure: Number; unit: participants
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Number analyzed (Participants) | 24 | 9
participants
  Baseline through Week 48 | 17 | 3
  Week 48 through Week 96 | 4 | 1
  Baseline through Week 96 | 21 | 4

ADVERSE EVENTS:
Time Frame: Baseline through Week 96 (Randomized Phase), and Week 96 up to a maximum of 954 days (Extension Phase)
Description: Safety Analysis Set
Arm/Group | FTC/RPV/TDF | EFV/FTC/TDF
Serious Adverse Events (participants affected / at risk) | 36/394 | 48/392
Other Adverse Events (participants affected / at risk) | 300/394 | 322/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=394) | EFV/FTC/TDF (N=392)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Neurosyphilis (Infections and infestations) | 0 | 2
Ophthalmic herpes zoster (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Eye infection syphilitic (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1
Secondary syphilis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testicular germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 2 | 2
Suicide attempt (Psychiatric disorders) | 1 | 3
Major depression (Psychiatric disorders) | 2 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Delirium tremens (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Behcet's syndrome (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/RPV/TDF (N=394) | EFV/FTC/TDF (N=392)
Diarrhoea (Gastrointestinal disorders) | 69 | 78
Nausea (Gastrointestinal disorders) | 65 | 65
Vomiting (Gastrointestinal disorders) | 20 | 21
Flatulence (Gastrointestinal disorders) | 24 | 9
Fatigue (General disorders) | 42 | 54
Pyrexia (General disorders) | 16 | 22
Upper respiratory tract infection (Infections and infestations) | 57 | 72
Nasopharyngitis (Infections and infestations) | 33 | 39
Bronchitis (Infections and infestations) | 34 | 29
Sinusitis (Infections and infestations) | 28 | 19
Syphilis (Infections and infestations) | 26 | 18
Folliculitis (Infections and infestations) | 27 | 8
Decreased appetite (Metabolism and nutrition disorders) | 10 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 20 | 13
Dizziness (Nervous system disorders) | 27 | 90
Headache (Nervous system disorders) | 56 | 61
Somnolence (Nervous system disorders) | 9 | 30
Abnormal dreams (Psychiatric disorders) | 23 | 101
Insomnia (Psychiatric disorders) | 45 | 60
Depression (Psychiatric disorders) | 34 | 47
Anxiety (Psychiatric disorders) | 28 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 38 | 27
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Rash (Skin and subcutaneous tissue disorders) | 31 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years